CLINICAL TRIAL: NCT01433432
Title: Clinical Efficacy and Safety of Delayed Release 6-Mercaptopurine (DR-6MP) for Targeted Ileal Delivery in Patients With Moderately Active Crohn's Disease - Open Label Extension Study
Brief Title: Open Label Extension Study to Protocol C2/13/DR-6MP-02
Acronym: OLE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrew support for study due to reorganization and project prioritization
Sponsor: Teva GTC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2/13/DR-6MP-02 EXT
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purinethol (Active Comparator): Subjects who previously received 12 weeks of Purinethol (at 1-1.5 mg/kg)in the original study will now receive 80 mg DR-6MP (2 x 40 mg tablets) once dailyh, in the evening, for an additional 12 weeks
  Interventions: Drug: 80 mg DR-6MP
- Test Drug (Experimental): Subjects who previously received test drug (80 mg DR-6MP) for 12 weeks in the original study, will continue to receive 80 mg DR-6MP (2 x 40 mg tablets) once daily, in the evening, for an additional 12 weeks
  Interventions: Drug: 80 mg DR-6MP

INTERVENTIONS:
Drug: 80 mg DR-6MP — All subjects from the original study, Protocol C2/13/DR-6MP-02, whether they received test drug for 12 weeks or Purinethol for 12 weeks, will now receive an additional 12 weeks of 80 mg DR-6MP drug to be administered as 2 x 40 mg DR-6MP test tablets, once nightly, before bedtime.

SUMMARY:
The open label extension study (Protocol C2/13/DR-6MP-02 EXT) is designed to evaluate the clinical efficacy and safety of 80 mg DR-6MP test formulation for an additional 12 weeks in subjects who already completed 12 weeks of Protocol C2/13/DR-6MP-02. Crohn's disease (CD) therapy is aimed at reducing inflammation via induction of remission after a flare-up and maintenance of the remission for as long as possible. The questions being asked in this extension study are:

1. For subjects who received 80 mg DR-6MP for 12 weeks: Can the clinical efficacy and safety status achieved following 12 weeks of treatment be maintained or improved following an additional 12 weeks of DR-6MP treatment?
2. For subjects who received oral Purinethol (1-1.5 mg/kg daily) for 12 weeks: Can the clinical efficacy and safety at 12 weeks be maintained or improved following the introduction of 12 weeks of 80 mg DR-6MP treatment?

DETAILED DESCRIPTION:
By following the 2 groups of subjects, i.e, those who originally received the test formulation (80 mg DR-6MP) and are now continuing for another 12 weeks on test drug vs. those who received the reference drug (Purinethol, 1-1.5 mg/kg daily) and are now being introduced to 12 weeks of 80 mg DR6MP test drug, and monitoring the CDAI scores, immunology parameters (ex. ESR and CRP) and safety assessments (i.e., adverse events occurrences, weight changes, laboratory test results) and comparing to the parameters at extension study start, the study will effectively answer the following questions:

1. Does an additional 12 weeks of 80 mg DR6MP test drug treatment maintain or improve CDAI scores?
2. Is an additional 12 weeks of 80 mg DR6MP test drug treatment safer due to negligible drug availability systemically?
3. Can an additional 12 weeks of 80 mg DR6MP test drug treatment evoke a more effective immunological systemic response?
4. In the subset of subjects willing to undergo colonoscopy/ileoscopy, does an additional 12 weeks of 80 mg DR6MP test drug induce effective mucosal healing?

ELIGIBILITY:
Inclusion Criteria:

1. Male and (non-pregnant) female subjects, who completed Protocol C2/13/DR-6MP-02, aged 18-75 years (inclusive)with no serious adverse events or complications and with the consent of the PI
2. Study entry screening laboratory tests must meet the following criteria:

   WBC greater than or equal to 3000mm3 ALT, AST less than 2 x upper limit of normal Total and direct bilirubin less than 2 x upper limit of normal Note: induction study Protocol C2/13/DR6MP-02 Week 12 termination labs can serve as screening labs for the extension study provided that the subject enters the extension study within 2 weeks of completing the induction study. If the interval is longer, however, repeat screening labs must be conducted.
3. Subjects must agree not to be taking any treatment for Crohn's disease other than stable dose of 5-ASA, chronic antibiotics or low-dose oral steroids (prednisolone up to 15 mg daily; budesonide up to 6 mg daily) at extension study entry and throughout the study.
4. Subjects willing and able to provide written informed consent.

Exclusion Criteria:

1. Subjects with a body weight at extension study entry below 42.5 kg
2. Women who are pregnant or nursing at the time of extension study entry or who intend to be during the study period
3. Women of childbearing potential who do not practice an acceptable method of birth control [acceptable methods of birth control are: surgical sterilization, intrauterine devices, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy, a double-protection method (condom or diaphragm with spermicide) or abstinence]
4. Subjects with planned elective surgery or hospitalization during the course of the study (that may interfere with study compliance or outcome)
5. Subjects who will be unavailable for the duration of the trial, are unable to comply with the planned schedule of study visits, are likely to be noncompliant with the protocol, or who are felt to be unsuitable by the investigator for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Maintenance of or reduction in CDAI score | 12 weeks
  Maintenance of or reduction in CDAI score at week 12X (end of extension study) relative to extension study start

SECONDARY OUTCOMES:
Maintenance of or improvement in safety assessments | 12 weeks
  Evaluate and compare the incidence, frequency and severity of Adverse Events between the 2 groups (those who previously received 80 mg DR6MP and continue to receive it vs. those who previously received Purinethol (1-1.5 mg/kg) and are now introduced to 80 mg DR6MP) over 12 weeks.
  This includes all Adverse Events reported, as well as changes in body weight and changes in clinically significant laboratory values, specifically, WBC, ALT, AST, direct and total bilirubin.

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Ilan, MD, Principal Investigator — Hadassah Medical Organization; Eran Goldin, MD, Principal Investigator — Shaare Zedek Medical Center